CLINICAL TRIAL: NCT01586234
Title: Randomized Clinical Trial of OCT-guided DSAEK Graft Shaping and Smoothing
Brief Title: OCT-guided DSAEK Graft Shaping and Smoothing
Acronym: DSAEK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, Mark Terry, MD, Director of Cornea Services, Legacy Health System
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB#00006612 DSAEK
Record Dates: First submitted 2012-01-03; First posted 2012-04-26 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Fuchs' Endothelial Dystrophy
Keywords: Fuchs' endothelial dystrophy; DSAEK; Descemet's stripping automated endothelial keratoplasty
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DSAEK with graft shaping and smoothing (Experimental)
  Interventions: Procedure: DSAEK with graft shaping and smoothing
- Standard DSAEK (Active Comparator)
  Interventions: Procedure: Standard DSAEK

INTERVENTIONS:
Procedure: DSAEK with graft shaping and smoothing — 1. A 5mm incision will be made in the sclera (white portion) of the eye, approximately 1mm from the edge of the cornea
  2. The tissue on the underside of the cornea (endothelium) will be scraped away
  3. The graft from the donor cornea (previously smoothed with a laser) will be inserted through the incision and placed against the endothelium of the host cornea.
  Arms: DSAEK with graft shaping and smoothing
Procedure: Standard DSAEK — 1. A 5mm incision will be made in the sclera (white portion) of the eye, approximately 1mm from the edge of the cornea
  2. The tissue on the underside of the cornea (endothelium) will be scraped away
  3. The graft from the donor cornea will be inserted through the incision and placed against the endothelium of the host cornea.
  Arms: Standard DSAEK

SUMMARY:
The primary goal of this study is to determine if excimer laser smoothing of the cornea before Descemet's stripping automated endothelial keratoplasty (DSAEK)improves postoperative Best Spectacle Corrected Visual Acuity (BSCVA).

DETAILED DESCRIPTION:
Many surgeons are moving away from full thickness corneal transplantation (because of risks involving rejection, irregular astigmatism, and wound dehiscence) to partial thickness transplantations of either the anterior or posterior (endothelial) layers. However this technique is not without its drawbacks. DSAEK uses a mechanical microkeratome to cut the graft, but vision is limited by the roughness of the cut surface.

DSAEK can lead to significant refractive error due to the non-uniform shape of the microkeratome cut graft, and the roughness of the microkeratome cut surface limits vision to an average of 20/31. Optical coherence tomography (OCT)-guided laser shaping and smoothing may improve the refractive and visual outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adults with visual complaint and objective evidence of decreased vision due to corneal edema related to Fuchs' corneal endothelial dystrophy

Exclusion Criteria:

* Inability to give informed consent
* Inability to maintain stable fixation for OCT imaging
* Inability to commit to required visits to complete the study
* Eyes with concurrent cataract, retinal diseases, glaucoma, or other eye conditions that may limit the visual outcome after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08-31 (Actual); Study Completion 2014-08-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with better post-operative spectacle-corrected visual acuity when implant graft is smoothed with eximer laser versus no smoothing of the graft. | 24 months
  To determine whether OCT-guided excimer laser graft shaping improves postoperative visual acuity, including reduction of postoperative hyperopic shift and improvement of the predictability of postoperative refraction.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Terry, MD, Principal Investigator — Devers Eye Institute, Legacy Health
Locations (1):
- Devers Eye Insitute, Portland, Oregon, United States